CLINICAL TRIAL: NCT02995577
Title: Biomarkers for Feeding Intolerance in Infants With Complex Congenital Heart Defects Undergoing Single Ventricle Staged Palliation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Supriya Nair, Pediatric GI Fellow, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-16-0968
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Single Ventricle Physiology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Feeding tolerant: Patients that are able to reach 80-100% of full enteral feeds (whether fed by mouth or through a nasogastric tube) 7 days after the initiation of feeds. Patients will be excluded from this group if they are ever diagnosed with NEC at any time during this hospitalization.
  Interventions: Other: Feeding tolerant
- Feeding intolerant: Patients with GI symptoms (vomiting, abdominal distention, diarrhea, hematemesis, and/or hematochezia) that persist for 48 hours or longer while needing to be NPO, this patient is retrospectively categorized into the feeding intolerance group. Patients with feeding intolerance may also include infants that are made NPO, placed on bowel rest, and are started on antibiotics to rule out NEC, but are never diagnosed with NEC. Exclusion criteria include patients that are continued on antibiotics for greater than 48 hours due to diagnosed bacterial sepsis or diagnosed NEC, and those that have a positive blood, urine, or sputum culture.
  Interventions: Other: Feeding intolerant
- Necrotizing enterocolitis: Any infant that is diagnosed (radiographically, by Bell's criteria) with and treated for NEC.
  Interventions: Other: Necrotizing enterocolitis

INTERVENTIONS:
Other: Feeding tolerant
  Groups: Feeding tolerant
Other: Feeding intolerant
  Groups: Feeding intolerant
Other: Necrotizing enterocolitis
  Groups: Necrotizing enterocolitis

SUMMARY:
The purpose of this study is to investigates serum and stool biomarkers as predictors for post-operative feeding intolerance in infant patients with complex congenital heart defects who undergo single ventricle staged palliation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Full term gestational period (37 weeks gestation or greater)
* minimum of 2.5kg or greater body weight
* diagnosis of single ventricle physiology, or complex congenital cyanotic heart disease requiring staged palliation surgery in the form of Norwood-type procedure, systemic-to-pulmonary artery shunt, or pulmonary artery banding.

Exclusion Criteria:

* Have diseases affecting other organs,
* have major congenital anomalies such as Hirschsprung disease, imperforate anus, CHARGE syndrome, or VACTERL association.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be infants with complex congenital cyanotic heart disease requiring single ventricle staged palliation surgery at Children's Memorial Hermann Hospital (CMHH) at the Texas Medical Center. This will include neonates undergoing single ventricle staged palliation in the form of (a) Norwood-type procedure, (b) systemic-to-pulmonary artery shunt procedure, or (c) pulmonary artery banding.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Level of most abundant serum protein as determined by ELISA | baseline (3-5 days after initial cardiac surgery), within three weeks of the initial cardiac surgery
  We will select two proteins with top changes that are involved in the pathways for intestinal inflammation, and levels will be determined with either ELISA or other techniques that are available.
Level of second most abundant serum protein as determined by ELISA | baseline (3-5 days after initial cardiac surgery), within three weeks of the initial cardiac surgery
Level of stool biomarker interleukin-8 (IL-8) as determined by ELISA | baseline (3-5 days after initial cardiac surgery), within three weeks of the initial cardiac surgery
Level of stool biomarker calprotectin as determined by ELISA | baseline (3-5 days after initial cardiac surgery), within three weeks of the initial cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Nair, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States